CLINICAL TRIAL: NCT01394887
Title: Metformin Decreases Plasma Resistin Concentrations in Pediatric Patients With Impaired Glucose Tolerance: A Placebo-controlled Randomized Clinical Trial
Brief Title: Metformin & Inflammation in Pre-diabetic Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Niels Wacher, Head of Research Unit for Clinical Epidemiology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2002-718-0018
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2002-07

CONDITIONS: Glucose Intolerance; Inflammation; Diabetes
Keywords: Metformin, inflammation; resistin; impaired glucose tolerance; children
MeSH Terms: conditions — Glucose Intolerance; Inflammation; Diabetes Mellitus | interventions — Metformin; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin group (Active Comparator): this group received 850 mg metformin twice daily, along with recommended diet and exercise
  Interventions: Drug: Metformin
- placebo group (Placebo Comparator): This group received 850 mg of placebo twice daily, along with a recommended regimen of diet and exercise
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin — 850 mg of metformin twice daily over 12 weeks
  Other Names: Diet and physical activity
  Arms: metformin group
Drug: placebo — 850 mg gel capsules with starch (6.8 calories)as placebo
  Other Names: Diet and physical activity
  Arms: placebo group

SUMMARY:
Hypothesis. To determine the effect of metformin on the concentrations of resistin and other insulin resistance or inflammatory markers (C-reactive protein, cytokines, body weight, HbA1c, among others) in minors with glucose intolerance.

Children with glucose intolerance are given either metformin or placebo for 12 consecutive weeks.

High sensitivity C-reactive protein, TNF-alpha, IL-6, IL1-beta, resistin, leptin, adiponectin, glucose, insulin, HbA1c, lipid profile and transaminases are measured at the beginning and at the end of the period. Statistical analysis: t Student test; Friedman and Kruskal Wallis test are used. Variables are adjusted for: sex, age, baseline BMI and percentage weight change.

DETAILED DESCRIPTION:
Experimental, double-blind, randomized, prospective, placebo-controlled study. Patients aged 4-17 years old are selected from the endocrine outpatient clinic of the Hospital de Pediatria del CMN "Siglo XXI", and both patients and parents sign informed consent. They are scheduled for a fasting oral glucose tolerance test (OGTT) with 1.75 mg/kg of oral glucose. A blood sample is taken from antecubital vein at baseline and 120 minutes.

A high carbohydrate diet is indicated for 3 days prior to the test. All patients diagnosed with glucose intolerance are invited to participate. All followed an aerobic program of 30 to 45 minutes every day, an isocaloric diet from the moment of inclusion throughout the study period, in order to decrease the effect of nutrition modification in the metabolic and vascular parameters. A complete medical history is taken, recording family background of diabetes plus blood pressure, heart rate and Tanner stage13. Age, body weight, height, waist circumference are measured and recorded in percentile according to age and gender, and the body mass index is calculated (kg/m2), and recorded in percentile according to reference values of the Center for the Disease Control, Atlanta, GA14. Subjects are randomized for metformin or placebo. Both metformin and placebo are placed in capsules with gelatin to blind their aspect. Treatments are administered during 3 months. Children are evaluated monthly, measuring transaminases, glucose, creatinine, and uric acid. Measurements of C reactive protein, cytokines, adipokines, insulin concentrations, HbA1c levels and lipid profile are made at the beginning and end of the study. Insulin resistance was assayed by HOMA-IR index. Beta cell function is determined by using HOMA-β. These are complemented with an evaluation of diet, physical activity, and physical examination.

Treatment assignment: Two groups are formed, randomly assigned using a table of random numbers previously designed with the Epistat statistic package (Round Rock, Texas). When the screening finished, every child receives a consecutive number. This number corresponds to an envelope with a card identifying his/her medication flasks, containing 60 tablets of 850 mg or placebo. The content of the capsules is not identified, so both the physician and the patient are blinded. A blinded member of the study prepared the flasks and labeled them.

Participants take the capsules twice daily, at breakfast and dinner. They are instructed to take medication with meals in order to decrease the possibility of adverse effects (nausea, meteorism, diarrhea), which are checked during every visit. Hepatic function is monitored during the study.

FPG, total cholesterol, HDL-cholesterol, triglycerides, liver function tests and creatinine are measured using the Synchron CX analyzer (Beckman Systems, Fullerton CA), according to the standard protocols. The coefficients of variation for cholesterol and HDL-cholesterol are 3.3% and 2.5% respectively. Plasma leptin, adiponectin and insulin concentrations are measured in duplicate by radioinmmunoassay (Linco Research Inc, St Charles, MO). HbA1c is determined in whole blood using ion exchange high performance liquid chromatography (normal range 4-6). Plasma resistin is measured using Human Resistin Elisa Kit (PeproTech, Rock Hill, NJ, USA) read by Multiscan EX, Lab Systems, USA). Plasma IL-6, IL1-b, TNF-α concentrations are determined by ELISA using Quantike HS Human Immunoassay Kits (R&D Systems, Minneapolis, MN, USA), plasma C-reactive protein (hs-CRP) is measured using a highly sensitive human CRP ELISA Kit (Alpha diagnostic international, San Antonio, TX, USA ) according to the manufacturer's instructions and are read by an ELISA reader (Sunrise, Tecan USA, Durham NC,USA).

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with glucose intolerance per ADA criteria,
* free of acute or chronic inflammatory processes 3 months prior to recruitment,
* 4-17 years of age

Exclusion Criteria:

* previous personal history of diabetes or demonstrating diabetes in OGTT curve,
* chronic renal disease or serum creatinine over 1.4 mg/dl (females) or 1.5 (males),
* active hepatic disease,
* smoking,
* primary dislipidemia,
* heart problems,
* steroids,
* chronic metabolic acidosis,
* receiving anti-hypertensive or hypolipemia or hypoglucemia medications

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2002-07; Primary Completion 2003-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
presence of inflammation | 1 year
  to determine the efficacy of metformin in avoiding deterioration of glucose intolerance to type 2 diabetes, as measured by inflammation through various recognized inflammation markers

SECONDARY OUTCOMES:
presence of type 2 diabetes | 10 years
  to determine the efficacy of metformin in avoiding deterioration of glucose intolerance to type 2 diabetes, as measured by inflammation through various recognized inflammation markers

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Wacher, MD, Study Director — Supervisor Clinical Research
Locations (1):
- Endocrine Outpatient Clinic of the Hospital de Pediatria del CMN "Siglo XXI", Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Gomez-Diaz RA, Talavera JO, Pool EC, Ortiz-Navarrete FV, Solorzano-Santos F, Mondragon-Gonzalez R, Valladares-Salgado A, Cruz M, Aguilar-Salinas CA, Wacher NH. Metformin decreases plasma resistin concentrations in pediatric patients with impaired glucose tolerance: a placebo-controlled randomized clinical trial. Metabolism. 2012 Sep;61(9):1247-55. doi: 10.1016/j.metabol.2012.02.003. Epub 2012 Mar 17. PMID 22424822